CLINICAL TRIAL: NCT01840189
Title: Continuous Subcutaneous Hydrocortisone Infusion In Addison's Disease and Type 1 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012/2218; 2012/005516-26 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2016-12

CONDITIONS: Addison Disease; Type 1 Diabetes
Keywords: Addison disease; Type 1 diabetes; treatment
MeSH Terms: conditions — Addison Disease; Diabetes Mellitus, Type 1 | interventions — Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cortef (Active Comparator): Treatment A is oral hydrocortisone replacement( Cortef 5 mg)with weight-adjusted doses as suggested by Mah et al , will take 2 months
  Interventions: Other: Solu-cortef
- Solu-cortef (Active Comparator): This is the treatment B by continuous subcutaneous hydrocortisone infusion. Solu-cortef infusion will be given as Solu-Cortef Act-o-Vial 50mg/ml, , produced by Pfizer. Pump designed for subcutaneous insulin infusion can be used for subcutaneous administration.
  Interventions: Other: Cortef

INTERVENTIONS:
Other: Cortef — Treatment A is oral hydrocortisone replacement ( Cortef 5 mg) administered according to weight-adjusted doses for 2 months
  Arms: Solu-cortef
Other: Solu-cortef — Treatment B is continuous subcutaneous hydrocortisone infusion with the initial standard dose of 10mg/m2/24hrs. Body surface area will be calculated according to the nomogram from the formula of Du Bois and Du Bois.
  This part of the study will take 2 months.
  Arms: Cortef

SUMMARY:
The conventional glucocorticoid replacement therapy in primary adrenal insufficiency (Addison's disease) renders the cortisol levels unphysiological, which may cause symptoms and long-term complications.

The majority of Addison's patients have other organ-specific autoimmune disease, which poses challenges to the replacement therapy. Of particular interest is the combination of Addison's disease and type 1 diabetes, since cortisol affects glucose homeostasis. The clinical experience is that this subgroup of patients is difficult to treat, but very little research has been done to understand and improve their situation.

Glucocorticoid replacement is technically feasible by continuous subcutaneous hydrocortisone infusion, and can mimic the normal diurnal cortisol rhythm. This pilot study aims to further evaluate continuous subcutaneous hydrocortisone infusion treatment in terms of metabolic effects especially glycemic control in patients with the combination of Addison's disease and type 1 diabetes in an 5 months cross-over design open clinical pilot study.

DETAILED DESCRIPTION:
Treatment of Addison's disease includes glucocorticoid and mineralocorticoid replacement. Despite optimized therapy with these steroids, many patients suffer from impaired quality of life and increased mortality. The etiology of the premature death is complicated and may include a combination of inadequate treatment of adrenal crisis, patient non-compliance, and undetected hypoglycemia, in addition to being associated with increased cardiovascular, malignant, and infectious disease deaths. The relative risk of death for patients with Type 1 Diabetes is 3.8 in Sweden. Having Type 1 diabetes and Addison's disease significantly increased the risk of death when compared with having adrenal insufficiency alone. The risk for premature death in patients with the combination of Type 1 diabetes and Addison's disease has not been extensively studied and appears to contribute to a small portion of the increased mortality seen in patients with Addison's disease.

Cortisol has particularly potent effects on blood glucose levels, otherwise Addison's disease affects the production of cortisol, an important counterregulatory hormone for hypoglycaemia. Lack of cortisol might increase the risk of hypoglycemic episodes, whereas over-replacement might cause hyperglycemia. Because steroid replacement may cause significant insulin resistance, it is challenging to adjust insulin doses to maintain optimal glycemic control. Little is known about the effects of unphysiological glucocorticoid replacement therapy on glucose and lipid metabolism, but there has been concern about long-term metabolic consequence. Current glucocorticoid replacement results in large fluctuations in the cortisol levels directly influencing glucose homeostasis and, consequently, making accompanying insulin treatment difficult to manage. Different types, regimens and doses of glucocorticoids are now used in adrenal insufficiency, but none approximate the physiological rhythm. Hydrocortisone administration via a subcutaneous pump is a novel strategy that restores circadian cortisol rhythm in most patients.

The study will be open-labelled, cross-over designed, with comparison of two glucocorticoid replacement modalities to glycemic events in randomised order within each patient, as illustrated in figure.

Treatment A is optimised oral hydrocortisone ( Cortef 5 mg) replacement according to Mah et al, and treatment B is continuous subcutaneous hydrocortisone infusion therapy. The patients will be assigned a participation number and randomised to any of two treatment sequences (A-B or B-A). Should the need for an extra glucocorticoid dose occur (intercurrent illness, exercises) during the study, for safety reasons, the patients should administer their previous glucocorticoid and insulin replacement. If the dose of insulin is changed, new testing by self-monitoring of blood glucose and continuous glucose monitor system should be done.

The period of dose adjustments for insulin treatment during both glucocorticoids replacement modalities will take 2 weeks for each and 6 weeks assessment of glycemic control by continuous glucose monitor system, followed by a minimal of one month during which the patients use their previous glucocorticoid replacement and previous insulin therapy (wash-out period).

Patients will be educated in groups, and dose adjustments will be co-ordinated with regular visits at the outpatient clinic/telephone consultation combined with laboratory analyses. After the principal study period participants will be offered a 3 months' continuous subcutaneous hydrocortisone infusion treatment extension period. Infusion gear and Solu-Cortef 50mg/ml infusate will be refunded over the study budget. Hydrocortisone infusion will be given as Solu-Cortef Act-o-Vial 50mg/ml produced by Pfizer. Pump designed for subcutaneous insulin infusion can be used for subcutaneous administration.

glucose levels are stable.

Withdrawal criteria/Adverse Events The patient is free to withdraw at any time. If a patient is having major difficulties managing the infusion pump/equipment/continuous glucose monitor after thorough education and instructions, the investigator will consider withdrawal. In the best interest of the patient, the investigator and the sponsor can decide to withdraw the patient from the study. Compliance of the patients will be checked according to the report from remote control - Patients Diabetes Manager and continuous glucose monitor. Unfortunately, there are available no methods how to follow up the compliance to the oral treatment. If a patient develops conditions meeting the exclusion criteria, the patient will be withdrawn from the study. In case of serious adverse events the patient may be withdrawn from the study.

Any adverse event will be registered and reported to the Norwegian and Swedish Medicines Agency. Any serious adverse events will be reported within 15 days, and in case of lethal or life threatening events immediately. The patients will report any problems or discomfort in the patient diary, any need for extra doses with glucocorticoids will also be documented there. In addition, we ask them to contact the study group directly in case of problems/adverse events between consultations.

The study documentation and research date will be stored 15 years after the termination of the study. After the termination of the study we will notify ethical committee by 90 days and the final report will be prepared and delivered to ethical committee. If needed to terminate the study earlier, we will notify the ethical committee by 15 days.

Statistical considerations The studies are academic, investigator-driven pilot studies, limited in number by expensive techniques and rare diseases.

ELIGIBILITY:
Inclusion Criteria:

- primary Addison's disease in combination with long-standing Type 1 diabetes

Exclusion Criteria:

* cardiovascular disease
* active malignant disease
* pregnant women
* pharmacological treatment with glucocorticoids or drugs that interfere with cortisol metabolism (antiepileptics, rifampicin, St. Johns war, estrogens)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
nocturnal hypoglycemic events | 4 months
  severe hypoglycemia (needs for another person's assistance, blood glucose ≤ 3.1 mmol ⁄ L or prompt recovery after oral carbohydrate, i.v glucose or glucagon administration) and insulin requirement

SECONDARY OUTCOMES:
o Nocturnal glycemic variability | 4 months
  monitored by continuous glucose monitor system
hormone and metabolic profile | 4 months
  * Hormone levels : insulin like growth factor 1, growth hormone
  * Steroid metabolism: adrenocorticotropic hormone , cortisol
  * Metabolic profile: fructosamine, HBA1C, lipid levels, C reactive protein , homeostasis model assessment index
o Subjective health status | 4 months
  Self administration of questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Løvås, MD, PhD, Study Director — Haukeland University Hospital; Katerina Simunkova, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospiatl, Bergen, Norway

REFERENCES:
- [Background] Van den Driessche A, Eenkhoorn V, Van Gaal L, De Block C. Type 1 diabetes and autoimmune polyglandular syndrome: a clinical review. Neth J Med. 2009 Dec;67(11):376-87. PMID 20009114
- [Background] Barker JM. Compounding risk for hypoglycemia: type 1 diabetes and Addison's disease. Diabetes Technol Ther. 2012 May;14(5):383-5. doi: 10.1089/dia.2012.0043. Epub 2012 Apr 16. No abstract available. PMID 22506859
- [Background] Berger B, Stenstrom G, Sundkvist G. Incidence, prevalence, and mortality of diabetes in a large population. A report from the Skaraborg Diabetes Registry. Diabetes Care. 1999 May;22(5):773-8. doi: 10.2337/diacare.22.5.773. PMID 10332680
- [Background] Bergthorsdottir R, Leonsson-Zachrisson M, Oden A, Johannsson G. Premature mortality in patients with Addison's disease: a population-based study. J Clin Endocrinol Metab. 2006 Dec;91(12):4849-53. doi: 10.1210/jc.2006-0076. Epub 2006 Sep 12. PMID 16968806
- [Background] Elbelt U, Hahner S, Allolio B. Altered insulin requirement in patients with type 1 diabetes and primary adrenal insufficiency receiving standard glucocorticoid replacement therapy. Eur J Endocrinol. 2009 Jun;160(6):919-24. doi: 10.1530/EJE-08-1003. Epub 2009 Mar 9. PMID 19273569
- [Background] Johannsson G, Nilsson AG, Bergthorsdottir R, Burman P, Dahlqvist P, Ekman B, Engstrom BE, Olsson T, Ragnarsson O, Ryberg M, Wahlberg J, Biller BM, Monson JP, Stewart PM, Lennernas H, Skrtic S. Improved cortisol exposure-time profile and outcome in patients with adrenal insufficiency: a prospective randomized trial of a novel hydrocortisone dual-release formulation. J Clin Endocrinol Metab. 2012 Feb;97(2):473-81. doi: 10.1210/jc.2011-1926. Epub 2011 Nov 23. PMID 22112807
- [Background] Lovas K, Husebye ES. Continuous subcutaneous hydrocortisone infusion in Addison's disease. Eur J Endocrinol. 2007 Jul;157(1):109-12. doi: 10.1530/EJE-07-0052. PMID 17609409
- [Background] Bryan SM, Honour JW, Hindmarsh PC. Management of altered hydrocortisone pharmacokinetics in a boy with congenital adrenal hyperplasia using a continuous subcutaneous hydrocortisone infusion. J Clin Endocrinol Metab. 2009 Sep;94(9):3477-80. doi: 10.1210/jc.2009-0630. Epub 2009 Jun 30. PMID 19567522
- [Background] Mah PM, Jenkins RC, Rostami-Hodjegan A, Newell-Price J, Doane A, Ibbotson V, Tucker GT, Ross RJ. Weight-related dosing, timing and monitoring hydrocortisone replacement therapy in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2004 Sep;61(3):367-75. doi: 10.1111/j.1365-2265.2004.02106.x. PMID 15355454
- See also: Endocrine Society — http://www.ese-hormones.org